CLINICAL TRIAL: NCT05505396
Title: Hyperglycaemia and Hyperlactataemia in Patients With Severe Acute Brain Injury in the Intensive Care Unit - a Prospective, Observational Cohort Study
Brief Title: Hyperglycaemia and Hyperlactataemia in Patients With Severe Acute Brain Injury
Acronym: BRAIN-GLULAC
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Alexandra Vassilieva, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: P-2022-321
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Acute Brain Injury; Hyperglycemia; Hyperlactatemia
MeSH Terms: conditions — Brain Injuries; Hyperglycemia; Hyperlactatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Sampling of blood and cerebrospinal fluid — Blood HbA1c, insulin, C-peptide and IL-6 measured at admission. Glucose and lactate measured every 4 hours during intensive care stay. Daily sampling of CSV analysed for glucose and lactate in patients with EVD.

SUMMARY:
This is an observational study of patients with severe acute brain injury, which aims to characterize the development of hyperglycaemia and hyperlactataemia and the influence of these markers on clinical outcome.

Additionally, in a subgroup of patients undergoing advanced multimodal neuromonitoring on either clinical or research indication, the relationship between hyperglycaemia and brain glucose levels as well as systemic and microdialysis lactate will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to the neurointensive care unit at Rigshospitalet
* Diagnosis of acute brain injury categorised as TBI, SAH, ICH, ischaemic stroke, or other conditions

Exclusion Criteria:

* Brain death before inclusion
* Closest relatives do not understand written and spoken Danish or English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include all patients with severe acute brain injury, admitted to the neuro intensive care department at Rigshospitalet, Denmark. Mainly, it will be patients with TBI, SAH, ICH or acute ischaemic stroke.
Sampling Method: Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Functional outcome at 6 months as evaluated by the modified Rankin Scale. | 6 months after admission.
  Modified Rankin Scale ranges from 0-6, where 0 is the best and 6 is the worst outcome.

SECONDARY OUTCOMES:
All-cause mortality at 6 months (dichotomous). | 6 months after admission.
Length of stay in the neuro-ICU (continuous). | Day of discharge, typically 1-30 days after admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neuroanesthesiology and Neurointensive Care, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
IPD will only be shared with a data sharing agreement.